CLINICAL TRIAL: NCT06542029
Title: Groups 4 Health (Ryhmät Kuntoon) for Mental Well-being: a Feasibility and Controlled Effectiveness Study At the University of Helsinki
Brief Title: Interventions for the Wellbeing of Students At the University of Helsinki
Acronym: INSIGHT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: Strategic Research Council, Finland (Unknown); University of Eastern Finland (Other); Finnish Institute for Health and Welfare (Other Government)
Responsible Party: Principal Investigator, Jari Lahti, Professor, University of Helsinki
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SRC 352700
Record Dates: First submitted 2024-02-02; First posted 2024-08-07 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Well-Being, Psychological
Keywords: University Students; Group Intervention; Mental Health; Loneliness; Social Isolation; Anxiety; Depression; Social Anxiety; Social Cohesion; Equality; Inclusion; Motivation; Controlled study; Groups 4 Health; Adherence; Acceptance and Commitment Therapy
MeSH Terms: conditions — Psychological Well-Being; Social Isolation; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: This study is a parallel-arm non-randomized controlled clinical trial. The participants are assigned to the different intervention arms based on their preference (the students can sign up for an intervention of their choosing).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Groups 4 Health (G4H) (Experimental): Groups 4 Health (G4H, "Ryhmät kuntoon") intervention is administered in this arm.
  Interventions: Behavioral: Groups 4 Health (G4H)
- The study psychologists' group intervention (Active Comparator): The study psychologists' group intervention is administered in this arm.
  Interventions: Behavioral: The study psychologists' group intervention
- Towards better well-being and studying -online course (Active Comparator): Online course for students' well-being and studying ("Kohti parempaa opiskelua") is administered in this arm.
  Interventions: Behavioral: Towards better well-being and studying -online course
- No intervention control group (No Intervention): The no intervention control group consists of students who are not attending any active interventions for mental well-being or promotion of studying skills.

INTERVENTIONS:
Behavioral: Groups 4 Health (G4H) — Groups 4 Health, G4H, ("Ryhmät kuntoon") at the University of Helsinki is a manualized group intervention for the students that focuses on social connectedness and aims at improving general health and life satisfaction. G4H groups are facilitated by two psychology MA students (or licensed psychologists) carefully trained for the intervention and mentored by experienced clinical psychologists. G4H consists of five 90 minutes sessions that aim to give participants the knowledge and skills they need to effectively manage their social group memberships and identities. Each session contains exercises and discussions described in the G4H workbook that target different aspects of group life identified within the social identity model of identity change and put the Social Identity Approach to Health -model to practice. Students earn 2 ECTS (European Credit Transfer and Accumulation System) credits for completing the intervention.
  Other Names: Ryhmät kuntoon
  Arms: Groups 4 Health (G4H)
Behavioral: The study psychologists' group intervention — University of Helsinki study psychology team organizes group interventions for various challenges of studying for bachelor's and master's students. These groups offer client-centered peer support facilitated by one to two study psychologists. Recurring themes in the groups include: challenges in attentiveness, independent studying, and scientific writing, as well as support for re-entering the studies after a break. The approach in the different thematic groups is largely similar: short presentations, group discussions and practices. These groups have been implemented as both face-to-face and remote meetings. One group typically lasts for a study period and comprises five to six 90 minutes sessions. Typical group size is six to 12 students.
  Arms: The study psychologists' group intervention
Behavioral: Towards better well-being and studying -online course — Towards better well-being and studying -online course ("Kohti parempaa opiskelua") is an optional, seven-week online course that aims to foster university students' well-being and study skills. It is available for all University of Helsinki students. The course is based on principles of Acceptance and Commitment therapy and aims to support the development of psychological flexibility. The course takes place in Moodle platform and the students earn 3 ECTS credits for completing it. This course progresses week by week and has six central themes which include individual work in practicing psychological flexibility skills as well as study skills on a weekly basis and weekly group discussion.
  Arms: Towards better well-being and studying -online course

SUMMARY:
The psychological, social, and health consequences of psychological ill-being, particularly loneliness, are well-documented among students, which underlines the importance of providing adequate support. Groups 4 Health (G4H) is a promising psychosocial group intervention focused on improving well-being by supporting social connectedness and belonging.

In earlier Australian studies G4H has decreased loneliness and social anxiety and increased group memberships significantly more than treatment as usual. When compared to cognitive behavioral therapy G4H has showed continued reduction in the participants' loneliness at the end of the intervention period and in the follow-up.

Research on the G4H intervention's effectiveness outside Australia and research on the intervention's cost-effectiveness is lacking. Therefore, this clinical study investigates the feasibility, effectiveness, and cost-effectiveness of the G4H among the University of Helsinki students in Finland.

The effectiveness and cost-effectiveness of the G4H will be compared to two other active intervention groups: the well-being groups facilitated by the study psychologists at the University of Helsinki and an online course for students' well-being. Effectiveness will also be compared to students who do not participate in any well-being courses or interventions. The investigators hypothesize that all the active intervention groups promote student well-being.

Questionnaires and University of Helsinki registry data will be gathered before and after the interventions to evaluate the effectiveness and cost-effectiveness of the interventions. The factors that influence the intervention's effectiveness and cost-effectiveness will also be studied.

In addition to these research questions, qualitative methods are used to explore the challenges and possibilities identified in the G4H-intervention regarding inclusion and equality.

DETAILED DESCRIPTION:
Groups for health (G4H) is a manualized brief intervention based on social identity theory aiming to improve mental well-being by promoting social connectedness and belonging as well as reducing loneliness by building the participants' social identity capital in the context of group experience.

The Effectiveness of the G4H intervention has been studied in two Australian randomized controlled trials (RCT) as well as in one Australian controlled experiment. The RCT studies showed that G4H decreased loneliness and social anxiety and increased group memberships significantly more than treatment as usual and that in comparison with cognitive-behavioral therapy (CBT), both interventions reduced loneliness as effectively in the beginning of the intervention period, but the G4H group showed continued reduction in loneliness at the end of the intervention period and in the follow-up. Both interventions reduced depressive symptoms significantly and there were no differences between G4H and CBT. In all three controlled studies on the effects of G4H, inclusion criteria for the study were low mood and loneliness.

At present research on the effectiveness of G4H outside Australia is lacking and the cost-effectiveness of the G4H intervention or determinants of intervention effectiveness have not been evaluated. Consequently, this study focuses on the feasibility, effectiveness, and cost-effectiveness of the G4H among the University of Helsinki (UH) students in Finland. Moreover, students will not be excluded based on lack of loneliness or symptoms of depression.

The participants are students at the UH who have either; A) applied for three brief interventions for students' well-being: "Ryhmät kuntoon" -course (G4H at the UH), groups facilitated by the study psychologists, or online course for students' well-being (active intervention groups), or B) students who are not attending to any active interventions for mental well-being or promotion of studying skills (no-intervention control group). The students will be recruited for the active intervention groups and no-intervention group by email, website, and social media advertisements circulated by the UH media and communications services, communications services at the faculties, student health services, and student organizations. The interventions will be organized at the UH and are free for the UH students.

Data on the outcome measures is collected before and during the intervention as well as in 1- and 3-months follow-ups. Appropriate statistical methods including linear mixed model analyses will be used to study the effectiveness of the G4H intervention.

In addition to the outcome measures, data on the participants' and facilitators' background will be collected. The participant background questionnaire is filled out before the intervention and it consists of information on age, gender, birth date, mother tongue, marital status, household composition, residential situation, employment status, education, income, subjective health, readiness to attend to the intervention, social support, academic skills, and situational intrinsic and extrinsic motivation. Data gathered from UH registries include information on study rights (faculty, degree programs, fields of study) and their starting years, on active and passive registration, completed degrees, and information on learning and studies, such as approaches to learning, experiences of the teaching-learning environment, stress, and experiences of study-related burnout during studies and work during studies (HowULearn and HowUStudy questionnaires). This data is gathered to account for these factors in the statistical analyses and to analyze if these factors influence the effectiveness and cost-effectiveness of the intervention.

To investigate how facilitators' individual professional and personal characteristics may predict intervention process and effectiveness, G4H facilitators will fill self-report measures both before and during the interventions. Before initiating the intervention, facilitators will fill questionnaires related to personality traits (Extra-Short Five questionnaire), attachment style (Experiences in Close Relationships -questionnaire), and self-experiences in close personal relationships (Trainee Background Information Form). After the week 3 session, the facilitators' experiences of their current skillfulness, difficulties, and emotions in group work is measured based on an abbreviated version of the self-reported Trainee Current Practice Report. In addition, the facilitators' experiences of the group working alliance will be surveyed, based on a modified version of the Therapist Working Alliance Inventory Short Form.

In the collection of the quantitative data, both paper-and-pencil and electronic versions of the questionnaires will be used. Those in the active intervention groups will fill in the data as part of the sessions during the interventions or in the frequency of the sessions if the questionnaires are provided electronically and those in the no-intervention group will fill-in the questionnaires based on the email reminders of the electronic data collection system (time interval between reminders resembling interval between sessions in the active intervention groups). Data is collected before the intervention, during the intervention (week 3), immediately after the intervention and in one- and three-months follow-ups.

In addition to the quantitative data collection the investigators will explore the challenges and possibilities identified in the G4H-intervention regarding inclusion and equality. Three methods of data collection are used: 1) participant observations, 2) interviews with G4H participants and facilitators and 3) focus groups with young people who belong to minorities. In this sub-study, the aim is to examine challenges and possibilities identified in the G4H-intervention regarding inclusion and equality and whether G4H promotes long-term inclusion and equality among the participants.

Participant observations are conducted in the meetings of the G4H group and interviews are conducted with a subset of facilitators and intervention participants in the end of the intervention period. The follow-up interviews will be conducted 6 months, 12 months and 3 years after the first interview. The facilitators and participants of G4H will be mailed information about the study and an informed consent will be acquired before the first session. The participant observation focuses on the interaction in the groups and the experiences of facilitators and participants, in order to gain knowledge about how the groups work, what kinds of issues they deal with and especially how inclusion and equality are accomplished in the groups (are there minority participants, can participants influence the themes dealt with in the groups, or is inclusion and equality taken into account in some other ways in the groups). Following the ethnographic research tradition, the researcher takes part in the activities of the groups instead of observing them from the outside. Depending on their preferences, the study participants (both facilitators and participants in the groups) will be interviewed in a group, in pairs or individually, in facilities located outside the university (for example in a study room of a local library).

In addition, focus groups are arranged with young people belonging to minority groups with increased risk of marginalization or mental health problems. In the focus groups, young people are asked to comment on the design/description of G4H in terms of equality and inclusion, with the goal of enhancing inclusivity by listening to their views on the interventions and accumulation knowledge on the fit between the interventions and their specific needs. The focus groups target young people belonging to sexual and/or gender minorities, young people with immigrant background and young people with disabilities. These groups represent youth minorities with a high risk of loneliness. To date, research on their experiences of different services is lacking. All the interviews will be tape-recorded and later transcribed.

Written informed consent is gathered from all participants. The participants who have given their consent have the option to withdraw from the study at any point. Students who are currently undergoing other (mental health) treatment will not be interviewed to avoid causing them further stress.

ELIGIBILITY:
Inclusion criteria

* Adult (age 18 and above)
* Student in the University of Helsinki, Finland
* Able to speak/read Finnish, Swedish, or English

Exclusion criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-03-20 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Loneliness | 1) Before the intervention, 2) During the intervention (week 3), 3) immediately after the intervention, 4) one month follow-up, 5) three months follow-up
  Loneliness is measured with the 4 and 8-item short forms of the revised University of California, Los Angeles Loneliness Scale (ULS-4 and ULS-8, response options: 1=never, 2=rarely, 3=sometimes, 4=often, lower score means better outcome).
Depression | 1) Before the intervention, 3) immediately after the intervention 4) one month follow-up, 5) three months follow-up
  Symptoms of depression are assessed with the 9-item Patient Health Questionnaire (response options: 0=not at all, 1=several days, 2=more than half the days, 3=nearly every day, lower score means better outcome).

SECONDARY OUTCOMES:
Active group memberships | 1) Before the intervention, 3) immediately after the intervention 4) one month follow-up, 5) three months follow-up
  Multiple group memberships are assessed with the 4-item Exeter Identity Transition Scale (response options: 1 = strongly disagree, 7 = strongly agree, higher score means better outcome).
Mental well-being | 1) Before the intervention, 2) immediately after the intervention 3) one month follow-up, 4) three months follow-up
  Mental well-being is assessed with the 7-item Short Warwick-Edinburgh Mental Wellbeing Scale (response options: 1=not at all, 2=rarely, 3=occasionally, 4=often, 5=all the time, higher score means better outcome).
General well-being | 1) Before the intervention, 3) immediately after the intervention 4) one month follow-up, 5) three months follow-up
  General well-being is assessed with the 14-item General Population version of the Clinical Outcomes in Routine Evaluation (response options: 0=not at all, 1=only occasionally, 2=sometimes, 3=often, 4=most of/all of the time, lower score means better outcome).
Anxiety | 1) Before the intervention, 3) immediately after the intervention 4) one month follow-up, 5) three months follow-up
  Symptoms of anxiety are assessed with the 7-item Generalized Anxiety Disorder Questionnaire (response options: 0=not at all, 1=several days, 2=more than half the days, 3=nearly every day, lower score means better outcome).
Social anxiety | 1) Before the intervention, 3) immediately after the intervention 4) one month follow-up, 5) three months follow-u
  Social anxiety is assessed with the 3-item Mini Social Phobia Inventory (response options: 0=not at all, 1=several days, 2=more than half the days, 3=nearly every day, lower score means better outcome).
Health-related quality of life | 1) Before the intervention, 2) immediately after the intervention, 3) three months follow-up
  Health-related quality of life is measured with the Euro Quality of Life - 5 dimension - 5 level questionnaire (EQ-5D-5L). The measure has 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) comprising of five statements of which the respondent can choose the option that best describes their situation. Higher score means better outcome. This measure is used to calculate the cost-effectiveness of the interventions.
Use of social and health care services | 1) Before the intervention, 2) immediately after the intervention, 3) three months follow-up
  The use of social and health care services for mental health is measured with a self-report questionnaire (medications, health care appointments, hospitalization, counseling). The use of health care services will be monetarized by using Finnish national unit costs. This measure is used to calculate the cost-effectiveness of the interventions.
Time used by facilitators | Immediately after each intervention session, during 8 weeks
  The time used for planning, executing, and assessing the G4H sessions is reported by the facilitators. This measure is used to calculate the cost-effectiveness of the interventions.
Study credits | 1 year before the intervention, 1 year after the intervention
  Overall accumulated study credit data is gathered from the UH registries. These data will be used both as measures of effectiveness of the interventions and to account for the confounders in the statistical analyses.
Grade point average | 1 year before the intervention, 1 year after the intervention
  One year grade point average is gathered from the UH registries. These data will be used both as measures of effectiveness of the interventions and to account for the confounders in the statistical analyses.
Weighted grade point average | 1 year before the intervention, 1 year after the intervention
  Weighted grade point average is determined by the grades of each course weighted by the number of credits gained for it.

OTHER OUTCOMES:
Mood | 1) Before the intervention, 2) During the intervention (week 3), 3) immediately after the intervention, 4) one month follow-up, 5) three months follow-up
  Mood is measured with scale from 0 (extremely bad mood) to 7 (extremely good mood)
Identification with the intervention | During intervention (week 3)
  Identification with the intervention group is assessed with the Single-Item Social Identification -measure (response options: 1 = fully disagree, 7 = fully agree, higher score means better outcome).
Participant adherence | Immediately after each intervention session, during 8 weeks
  The number of participants consented vs the number of participants completing the intervention, attendance rate of individual sessions
Facilitator's fidelity to the manual | Immediately after each intervention session, during 8 weeks
  To monitor fidelity to the G4H manual, the facilitators of the G4H groups will complete a short checklist at the end of each session to determine compliance to the protocol.
Participants' Working alliance | During intervention (week 3)
  Participants' experience of working alliance is assessed with the 12-item Working Alliance Inventory Short and Revised (response options: 1 = never, 2 = rarely, 3 = occasionally, 4 = sometimes, 5 = often, 6 = very often, 7 = always, 3 subscales: goal, task, bond, higher score means better outcome)
Facilitators' Working alliance | During intervention (week 3)
  Facilitators' working alliance is assessed with an 18-item version of the Therapist Working Alliance Inventory Short Form (response options: 1 = never, 2 = rarely, 3 = occasionally, 4 = sometimes, 5 = often, 6 = very often, 7 = always, 3 subscales: goal, task, bond, higher score means better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Jari M Lahti, PhD, Principal Investigator — University of Helsinki
Locations (1):
- University of Helsinki, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Asikainen H, Katajavuori N. Development of a Web-Based Intervention Course to Promote Students' Well-Being and Studying in Universities: Protocol for an Experimental Study Design. JMIR Res Protoc. 2021 Mar 9;10(3):e23613. doi: 10.2196/23613. PMID 33687336
- [Background] Connor KM, Kobak KA, Churchill LE, Katzelnick D, Davidson JR. Mini-SPIN: A brief screening assessment for generalized social anxiety disorder. Depress Anxiety. 2001;14(2):137-40. doi: 10.1002/da.1055. PMID 11668666
- [Background] Cruwys T, Haslam C, Rathbone JA, Williams E, Haslam SA, Walter ZC. Groups 4 Health versus cognitive-behavioural therapy for depression and loneliness in young people: randomised phase 3 non-inferiority trial with 12-month follow-up. Br J Psychiatry. 2022 Mar;220(3):140-147. doi: 10.1192/bjp.2021.128. PMID 35049477
- [Background] Haslam C, Holme A, Haslam SA, Iyer A, Jetten J, Williams WH. Maintaining group memberships: social identity continuity predicts well-being after stroke. Neuropsychol Rehabil. 2008 Oct-Dec;18(5-6):671-91. doi: 10.1080/09602010701643449. PMID 18924001
- [Background] Haslam C, Cruwys T, Haslam SA, Dingle G, Chang MX. Groups 4 Health: Evidence that a social-identity intervention that builds and strengthens social group membership improves mental health. J Affect Disord. 2016 Apr;194:188-95. doi: 10.1016/j.jad.2016.01.010. Epub 2016 Jan 21. PMID 26828756
- [Background] Haslam C, Cruwys T, Chang MX, Bentley SV, Haslam SA, Dingle GA, Jetten J. GROUPS 4 HEALTH reduces loneliness and social anxiety in adults with psychological distress: Findings from a randomized controlled trial. J Consult Clin Psychol. 2019 Sep;87(9):787-801. doi: 10.1037/ccp0000427. PMID 31403815
- [Background] Hatcher RL, Lindqvist K, Falkenstrom F. Psychometric evaluation of the Working Alliance Inventory-Therapist version: Current and new short forms. Psychother Res. 2020 Jul;30(6):706-717. doi: 10.1080/10503307.2019.1677964. Epub 2019 Oct 17. PMID 31621525
- [Background] Hays RD, DiMatteo MR. A short-form measure of loneliness. J Pers Assess. 1987 Spring;51(1):69-81. doi: 10.1207/s15327752jpa5101_6. PMID 3572711
- [Background] Heinonen E, Orlinsky DE, Willutzki U, Ronnestad MH, Schroder T, Messina I, Loffler-Stastka H, Hartmann A. Psychotherapist Trainees' Quality of Life: Patterns and Correlates. Front Psychol. 2022 Mar 24;13:864691. doi: 10.3389/fpsyg.2022.864691. eCollection 2022. PMID 35401345
- [Background] Konstabel K, Lonnqvist JE, Leikas S, Garcia Velazquez R, Qin H, Verkasalo M, Walkowitz G. Measuring single constructs by single items: Constructing an even shorter version of the "Short Five" personality inventory. PLoS One. 2017 Aug 11;12(8):e0182714. doi: 10.1371/journal.pone.0182714. eCollection 2017. PMID 28800630
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] McKay MT, Andretta JR. Evidence for the Psychometric Validity, Internal Consistency and Measurement Invariance of Warwick Edinburgh Mental Well-being Scale Scores in Scottish and Irish Adolescents. Psychiatry Res. 2017 Sep;255:382-386. doi: 10.1016/j.psychres.2017.06.071. Epub 2017 Jun 21. PMID 28666244
- [Background] Postmes T, Haslam SA, Jans L. A single-item measure of social identification: reliability, validity, and utility. Br J Soc Psychol. 2013 Dec;52(4):597-617. doi: 10.1111/bjso.12006. Epub 2012 Nov 4. PMID 23121468
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Wei M, Russell DW, Mallinckrodt B, Vogel DL. The Experiences in Close Relationship Scale (ECR)-short form: reliability, validity, and factor structure. J Pers Assess. 2007 Apr;88(2):187-204. doi: 10.1080/00223890701268041. PMID 17437384
- [Background] Evans C, Connell J, Audin K, Sinclair A, Barkham M. Rationale and development of a general population well-being measure: Psychometric status of the GP-CORE in a student sample. Br J Guid Counc. 2005;33(2):153-73
- [Background] Guay F, Vallerand RJ, Blanchard C. On the assessment of situational intrinsic and extrinsic motivation: The Situational Motivation Scale (SIMS). Motiv Emot. 2000;24:175-213.
- [Background] Haslam C, Jetten J, Cruwys T, Dingle G, Haslam SA. The new psychology of health: Unlocking the social cure. Routledge; 2018.
- [Background] Hatcher RL, Gillaspy JA. Development and validation of a revised short version of the Working Alliance Inventory. Psychotherapy research. 2006;16(1):12-25.
- [Background] Iyer A, Jetten J, Tsivrikos D. Torn Between Identities: Predictors of Adjustment to Identity Change Self Continuity: Individual And Collective Perspectives. Psychology Press, New York, NY, US; 2008.
- [Background] Orlinsky DE, Strauss B, Rønnestad MH, Hill C, Castonguay L, Willutzki U, et al. A collaborative study of development in psychotherapy trainees. Psychotherapy Bulletin. 2015;50(4):21-5.
- [Background] Parpala A, Lindblom-Ylänne S. Using a research instrument for developing quality at the university. Quality in Higher Education. 2012;18(3):313-28.
- [Background] Sarason IG, Sarason BR, Shearin EN, Pierce GR. A brief measure of social support: Practical and theoretical implications. J Soc Pers Relat. 1987;4(4):497-510.
- [Background] Roberts RE, Lewinsohn PM, Seeley JR. A brief measure of loneliness suitable for use with adolescents. Psychol Rep. 1993 Jun;72(3 Pt 2):1379-91. doi: 10.2466/pr0.1993.72.3c.1379. PMID 8337350
- [Background] Russell D, Peplau LA, Cutrona CE. The revised UCLA Loneliness Scale: concurrent and discriminant validity evidence. J Pers Soc Psychol. 1980 Sep;39(3):472-80. doi: 10.1037//0022-3514.39.3.472. PMID 7431205